CLINICAL TRIAL: NCT04880590
Title: Sex or no Sex: That is the Question. Impact of Coital Sexual Intercourse on the Clinical Pregnancy Rate After Embryo Transfer.
Brief Title: Sex or no Sex: That is the Question.
Status: Recruiting | Type: Observational
Sponsor: Fundación Santiago Dexeus Font (Other)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Other Study IDs: FSD-SEX-2021-05
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Infertility, Female; Sexual Intercourse
MeSH Terms: conditions — Infertility, Female; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sex Intercourse: women with a heterosexual sexual relationship after embryo transfer
  Interventions: Other: Sex intercourse
- Non sex intercourse: women without a heterosexual sexual relationship after embryo transfer

INTERVENTIONS:
Other: Sex intercourse — A heterosexual sexual relationship
  Groups: Sex Intercourse

SUMMARY:
This study aims to evaluate the impact of sexual intercourse and orgasm in the 72 hrs following embryo transfer of blastocysts on the clinical pregnancy rate.

An impact on sexual activity and a decrease in the frequency of intercourse has been observed in infertile couples. In couples who undergo assisted reproductive technology (ART), sexual relations have an additional component that can condition them, such as the fear of influencing the outcome of the cycle.

The usual practice in ART cycles has evolved towards a preference for blastocyst-stage embryo transfer, both in fresh in vitro fertilization (IVF) cycles and in frozen embryo transfer (FET) cycles.

The investigators consider it important to elucidate whether coital intercourse after embryo transfer (ET) has an impact on the clinical pregnancy rate after the transfer of blastocyst-stage embryos.

DETAILED DESCRIPTION:
It is proposed to carry out an observational, prospective study, in which women with a heterosexual sexual relationship are included, who carry out an embryo transfer, in a FET cycle in the Dexeus Woman Reproduction Medicine Service and who agree to participate in the same.

ELIGIBILITY:
Inclusion Criteria:

* Women with a heterosexual sexual relationship
* That they carry out an embryo transfer, in a FET cycle

Exclusion Criteria:

* Exclusion criteria are not foreseen

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -After detailed oral and written information on the nature of the study, patients who meet the inclusion criteria will give their written consent. According to this consent, patients agree to have their data used and analyzed for the present study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6-7 weeks after transfer
  Clinical pregnancy rate measured by ultrasound with the presence of a positive fetal heartbeat

SECONDARY OUTCOMES:
Miscarriage rate | Until 13 weeks after embryo transfer procedure
  The loss of a pregnancy during the first 13 weeks of pregnancy
Live birth rate | Until 42 weeks after embryo transfer
  Number of live birth after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ata B, Abou-Setta AM, Seyhan A, Buckett W. Application of seminal plasma to female genital tract prior to embryo transfer in assisted reproductive technology cycles (IVF, ICSI and frozen embryo transfer). Cochrane Database Syst Rev. 2018 Feb 28;2(2):CD011809. doi: 10.1002/14651858.CD011809.pub2. PMID 29489026
- [Background] Fanchin R, Harmas A, Benaoudia F, Lundkvist U, Olivennes F, Frydman R. Microbial flora of the cervix assessed at the time of embryo transfer adversely affects in vitro fertilization outcome. Fertil Steril. 1998 Nov;70(5):866-70. doi: 10.1016/s0015-0282(98)00277-5. PMID 9806568
- [Background] Fanchin R, Righini C, Olivennes F, Taylor S, de Ziegler D, Frydman R. Uterine contractions at the time of embryo transfer alter pregnancy rates after in-vitro fertilization. Hum Reprod. 1998 Jul;13(7):1968-74. doi: 10.1093/humrep/13.7.1968. PMID 9740459
- [Background] Robertson SA, Prins JR, Sharkey DJ, Moldenhauer LM. Seminal fluid and the generation of regulatory T cells for embryo implantation. Am J Reprod Immunol. 2013 Apr;69(4):315-30. doi: 10.1111/aji.12107. PMID 23480148
- [Background] Stanford JB, Hansen JL, Willis SK, Hu N, Thomas A. Peri-implantation intercourse does not lower fecundability. Hum Reprod. 2020 Sep 1;35(9):2107-2112. doi: 10.1093/humrep/deaa156. PMID 32756956
- [Background] Tao P, Coates R, Maycock B. The impact of infertility on sexuality: A literature review. Australas Med J. 2011;4(11):620-7. doi: 10.4066/AMJ.20111055. Epub 2011 Nov 30. PMID 23386877
- [Background] Tremellen KP, Valbuena D, Landeras J, Ballesteros A, Martinez J, Mendoza S, Norman RJ, Robertson SA, Simon C. The effect of intercourse on pregnancy rates during assisted human reproduction. Hum Reprod. 2000 Dec;15(12):2653-8. doi: 10.1093/humrep/15.12.2653. PMID 11098040
- See also: Related Info — http://dexeus.com